CLINICAL TRIAL: NCT05993936
Title: The Effect Of E-Mobıle Traınıng Gıven In The Postnatal Perıod On Postnatal Comfort And Breastfeedıng Self-Effıcıency
Brief Title: The Effect Of E-Mobıle Traınıng Gıven Postnatal Perıod On Postnatal Comfort And Breastfeedıng Self-Effıcıency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, seda karaçay yıkar, Assistant professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 129
Record Dates: First submitted 2023-07-18; First posted 2023-08-15 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-08

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e mobile aplication (Experimental): Postpartum period mobile application; It is an application that is prepared according to the Android Operating System, can be downloaded free of charge from the Google Play Store, and offers training and live counseling services for women who have given birth.
  Interventions: Device: mobile application
- control (No Intervention): this group will only receive the standard care provided in the hospital. no intervention will be made

INTERVENTIONS:
Device: mobile application — A mobile application developed by researchers for the problems experienced in the postpartum period and downloaded from the play store.
  Arms: e mobile aplication

SUMMARY:
The period until the 42nd day after birth is called the postpartum period by the World Health Organization (WHO) Especially the first week of the postpartum period is the transition period both physiologically and psychologically, and the period when postpartum problems are at the highest level.This study was planned as a two-group control and e-mobile application in order to determine the effect of e-mobile training given in the postpartum period on postpartum comfort and breastfeeding self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

The ages of 18-35, Primiparous and multiparous pregnancy, Not clinical diagnosis of risky pregnancy, Able to understand and speak Turkish, Without communication difficulties and mental disabilities The mother and the baby have not developed any complications during pregnancy, delivery and postpartum period, Having a smart phone in the mobile application group, Those who have not attended childbirth preparation classes,

Exclusion Criteria:

* Preterm birth
* Postterm birth

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
mobile application aim 1 | postpartum 7th week
  Thanks to the mobile application, it is planned to develop women's breastfeeding self-efficacy. As the scale score increases, self-efficacy changes
mobile application aim 2 | postpartum 7th week]
  Thanks to the mobile application, it is expected that the postpartum comfort of women will changes. As the score obtained from the scale increases, the comfort changes

IPD SHARING:
Plan to Share IPD: No